CLINICAL TRIAL: NCT01090765
Title: A Phase I/II Study of TRC105 in Metastatic Castrate Resistant Prostate Cancer (CRPC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, William Dahut Jr., M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100062; 10-C-0062
Record Dates: First submitted 2010-03-19; First posted 2010-03-22 (Estimated); Results first posted 2015-02-13 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-04

CONDITIONS: Prostate Cancer; Metastatic Castrate Resistant Prostate Cancer
Keywords: Prostate; Tumor; Cancer; Hormone; Androgen; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — carotuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- TRC105 1 mg/kg every 2 weeks (Experimental): Intravenous infusion at 1 mg/kg every 2 weeks
  Interventions: Drug: TRC105
- TRC105 3 mg/kg every 2 weeks (Experimental): Intravenous infusion at 3 mg/kg every 2 weeks
  Interventions: Drug: TRC105
- TRC105 10 mg/kg every 2 weeks (Experimental): Intravenous infusion at 10 mg/kg every 2 weeks
  Interventions: Drug: TRC105
- TRC105 10 mg/kg weekly (Experimental): Intravenous infusion at 10 mg/kg weekly
  Interventions: Drug: TRC105
- TRC105 15 mg/kg every 2 weeks (Experimental): Intravenous infusion at 15 mg/kg every 2 weeks
  Interventions: Drug: TRC105
- TRC105 20 mg/kg every 2 weeks (Experimental): Intravenous infusion at 20 mg/kg every 2 weeks
  Interventions: Drug: TRC105

INTERVENTIONS:
Drug: TRC105

SUMMARY:
Background:

* Currently, there is no curative therapy for metastatic castrate-resistant prostate cancer (CRPC), a leading cause of death in men. However, researchers are exploring new treatments that involve drugs that prevent angiogenesis (the process by which new blood vessels are formed) and can slow or prevent tumor growth.
* TRC105 is an experimental drug that blocks angiogenesis, and has been studied for possible use in treating different kinds of cancer. However, it has not been validated to treat prostate cancer in general or CRPC in particular.

Objectives:

* To determine the effects of TRC105 as a treatment for CRPC
* To determine the safety and effectiveness of TRC105 in treating CRPC

Eligibility:

- Men at least 18 years of age who have been diagnosed with castrate-resistant prostate cancer for which existing treatments have not been effective.

Design:

* Eligible individuals will have a series of blood and other tests to determine their suitability for participating in the study.
* Participants will receive intravenous infusions of TRC105 in a 28-day treatment cycle. Participants will receive i.v. (intravenous) infusions of TRC105 every two weeks on days 1 and 15 of each 28-day cycle (cohorts 1, 2, 3, 5, and 6) and every week on days 1, 8, 15, and 22 of each 28 day cycle (cohort 4).
* Participants will receive different doses of TRC105 depending on when they enter the study, up to a maximum tolerated dose or optimum treatment dose.
* Frequent blood and urine tests will be performed during treatment, as well as other tests of cancer progression as directed by the study doctors. Participants will receive medicines to help prevent possible adverse side effects of TRC105, such as allergic reaction to the drug.
* Participants will continue treatment with TRC105 until they or the study team decides that the medication is not beneficial. No additional testing will be required unless participants discontinue the treatment because of side effects (which the study doctors will follow until the side effects are resolved).

DETAILED DESCRIPTION:
Background:

- Inhibition of angiogenesis has demonstrable antitumor efficacy against castrate-resistant prostate cancer (CRPC). TRC105 is a human/murine chimeric immunoglobulin heavy constant gamma 1 (IgG1) kappa monoclonal antibody that binds to human CD105 (endoglin), thus inhibiting angiogenesis and tumor growth. Data from an ongoing phase I clinical trial suggest that TRC105 is well tolerated with evidence of clinical efficacy in patients with metastatic CRPC.

Primary Objectives:

- Define the maximum tolerable dose (MTD) of TRC105 given every one to two weeks.

Secondary Objectives:

* Define the dose-limiting toxicities and toxicity profile of TRC105 given every one to two weeks
* Evaluate time to disease progression, overall response rate and overall survival.
* Describe the prostate specific antigen (PSA) response rate to therapy with TRC105
* Characterize the pharmacokinetics of TRC105
* Demonstrate a biologic effect of TRC105 in the patient and, when possible, on the tumor via laboratory evaluation of the molecular markers of angiogenesis before and after drug administration respectively

Eligibility:

* Progressive, castrate-resistant, metastatic adenocarcinoma of the prostate
* Eastern Cooperative Oncology Group (ECOG) less than or equal to 2

Design:

- An initial single-arm, phase I dose escalation study open to all patients with progressive metastatic CRPC. The study will evaluate patients in five cohorts of escalating dose levels. A maximum of 30 patients will be needed to complete the phase I evaluation.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patients must have histopathological confirmation of prostate cancer by the Laboratory of Pathology of the National Cancer Institute (NCI), Pathology Department of the National Naval Medical Center or Pathology Department of Walter Reed Army Medical Center prior to entering this study. Patients whose pathology specimens are no longer available may be enrolled in the trial if the patient has a clinical course consistent with prostate cancer and available documentation from an outside pathology laboratory of the diagnosis. In cases where original tissue blocks or archival biopsy material is available, efforts will be made to contact referring physicians and outside pathology departments to have the material forwarded to the research team for use in correlative studies.
  2. Patients must have metastatic progressive castrate-resistant prostate cancer defined as progressive disease (see below) despite surgical castration or ongoing use of gonadotropin-releasing hormone agonists with confirmed castrate levels of testosterone.

Criteria of progression for trial eligibility are defined from the Prostate Cancer Clinical Trials Working Group-2. Clinically progressive prostate cancer must be evidenced and documented by any of the following parameters:

1. Two consecutively rising prostate specific antigen (PSA) values at a minimum of 1-week intervals (2.0 ng/mL is the minimum starting value for PSA)
2. Appearance of one or more new lesion on bone scans
3. Progressive measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1

   Patients on flutamide for at least 6 months must have disease progression at least 4 weeks after withdrawal. Patients on bicalutamide or nilutamide for at least 6 months must have progression at least 6 weeks after withdrawal.

   All patients enrolled will be required to have measurable or non-measurable disease on imaging studies.

   4. Age greater than or equal to 18 years.

   5. Life expectancy of greater than 3 months.

   6. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.

   7. Patients must have normal organ and marrow function as defined below:
   * Absolute neutrophil count greater than or equal to 1,500/mcL
   * Platelets greater than or equal to 100,000/mcL
   * Total bilirubin less than or equal to 1.5 times upper normal limits or less than 3 mg/dl in subjects with Gilbert's Syndrome
   * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) less than or equal to 2.5 times upper limit of normal
   * Creatinine less than or equal to 1.5 times upper normal limits OR creatinine clearance greater than or equal to 40 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal, as calculated by the Cockcroft Gault formula.

     8. Patients must have recovered from any acute toxicity related to prior therapy, including surgery. Toxicity should be less than or equal to grade 1 or returned to baseline.

     9. All patients who have not undergone bilateral surgical castration must continue suppression of testosterone production by appropriate usage of gonadotropin releasing hormone (GnRH) agonists or antagonists.

     10. Patients must not have other invasive malignancies (within the past 2 years with the exception of non-melanoma skin cancers or non-invasive bladder cancer).

     11. Enrolled patients must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, the duration of study participation and 3 months after the end of the treatment.

     12. Patient must be able to understand and willing to sign a written informed consent document.

     13. Patients on a stable dose of steroids of 10 mg/day or less can continue on steroids if they are on peptic ulcer disease prophylaxis with an H2-blocker or proton pump inhibitor.

   EXCLUSION CRITERIA:
   1. Patients who have had chemotherapy, large field radiotherapy, or major surgery must wait 3 weeks prior to entering the study.
   2. Patients may not be receiving any agents not approved by the Food and Drug Administration (FDA) within the past 4 weeks.
   3. Patients with known brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
   4. Proteinuria, as demonstrated by a 24 hour protein of (Bullet) 2000 mg. Urine protein will be screened by urine protein-creatinine ratio (UPC). For UPC ratio > 1.0, a 24-hour urine protein will need to be obtained and the level should be < 2000 mg for patient enrollment.
   5. Uncontrolled intercurrent illness including, but not limited to, hypertension (systolic blood pressure (BP) > 160, diastolic BP > 100), ongoing or active systemic infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric illness/social situations that would limit compliance with study requirements.
   6. Thrombolytic or treatment-dose anticoagulant use within 10 days prior to first dose with TRC105.
   7. Hemorrhage within 30 days of dosing.
   8. History of peptic ulcer disease or gastritis within 6 months of TRC105 administration, unless patient has received adequate treatment for peptic ulcer disease and has evidence of complete resolution documented by esophagogastroduodenoscopy (EGD).
   9. Corrected QT interval (QTc) > 500 msec.
   10. Known human immunodeficiency virus (HIV)-positive patients are excluded.
   11. History of hypersensitivity reaction to human or mouse antibody products.
   12. Patients with a history of familial bleeding disorders.
   13. Patients with a history of hereditary hemorrhagic telangiectasia (Osler-Weber-Rendu syndrome).
   14. Use of non-steroidal anti-inflammatory drugs (NSAIDs) beginning 14 days prior to the first TRC105 dose, with the exception of aspirin when clinically indicated.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-02-23 (Actual); Primary Completion 2014-04-01 (Actual); Study Completion 2015-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William L Dahut, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Grossfeld GD, Stier DM, Flanders SC, Henning JM, Schonfeld W, Warolin K, Carroll PR. Use of second treatment following definitive local therapy for prostate cancer: data from the caPSURE database. J Urol. 1998 Oct;160(4):1398-404. PMID 9751363
- [Background] Figg WD, Feuer JA, Bauer KS. Management of hormone-sensitive metastatic prostate cancer. Update on hormonal therapy. Cancer Pract. 1997 Jul-Aug;5(4):258-63. No abstract available. PMID 9250085
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-C-0062.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study did not make it to the phase II (Arm 1-chemotherapy-naïve for metastatic disease (no prior antiangiogenic therapy) and Arm 2- post-docetaxel disease progression; evidence of disease progression despite prior docetaxel and bevacizumab) portion, thus no data is available for the phase II outcome measure "progression free survival".
Period: Overall Study
Arm/Group | TRC105 1 mg/kg Every 2 Weeks | TRC105 3 mg/kg Every 2 Weeks | TRC105 10 mg/kg Every 2 Weeks | TRC105 10 mg/kg Weekly | TRC105 15 mg/kg Every 2 Weeks | TRC105 20 mg/kg Every 2 Weeks
Started | 3 | 3 | 3 | 2 | 6 | 4
Completed | 3 | 3 | 3 | 1 | 4 | 3
Not Completed | 0 | 0 | 0 | 1 | 2 | 1
Not completed — Patient withdrew consent | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Developed a DVT, needed anticoagulation | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Vasovagal reaction with first infusion | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TRC105 1 mg/kg Every 2 Weeks | TRC105 3 mg/kg Every 2 Weeks | TRC105 10 mg/kg Every 2 Weeks | TRC105 10 mg/kg Weekly | TRC105 15 mg/kg Every 2 Weeks | TRC105 20 mg/kg Every 2 Weeks | Total
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 6 | 4 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 1 | 1 | 4 | 3 | 12
  >=65 years | 1 | 2 | 2 | 1 | 2 | 1 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (19.05) | 62.37 (9.01) | 66.53 (16.14) | 63.15 (4.45) | 65.83 (12.56) | 61.8 (7.56) | 64.32 (11.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 3 | 3 | 2 | 6 | 4 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 3 | 2 | 6 | 4 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 1 | 1 | 2 | 7
  White | 3 | 1 | 2 | 1 | 5 | 2 | 14
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 2 | 6 | 4 | 21

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD) of TRC105 Given Every Two Weeks.
Description: The MTD, to be administered in the phase II portion, is defined as the highest dose studied for which the incidence of dose limiting toxicity (DLT) was less than 33%. TRC105 was administered at 20 mg/kg intravenous every two weeks until MTD was achieved.
Time Frame: 6 months
Measure: Number; unit: mg/kg every 2 weeks
Arm/Group | TRC105 20 mg/kg Every 2 Weeks
Number analyzed (Participants) | 21
mg/kg every 2 weeks | 20

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: Date treatment consent signed to date off study, approximately 43 months, 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | TRC105 1 mg/kg Every 2 Weeks | TRC105 3 mg/kg Every 2 Weeks | TRC105 10 mg/kg Every 2 Weeks | TRC105 10 mg/kg Weekly | TRC105 15 mg/kg Every 2 Weeks | TRC105 20 mg/kg Every 2 Weeks
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 6 | 4
Participants | 3 | 3 | 3 | 2 | 5 | 4

3. Secondary Outcome: Dose Limiting Toxicity (DLT)
Description: Dose limiting toxicity is defined as any grade 3 or higher hematologic (excluding anemia) or non-hematologic toxicity considered to be possibly related to TRC105.
Time Frame: First 28 days on study
Measure: Count of Participants; unit: Participants
Arm/Group | TRC105 1 mg/kg Every 2 Weeks | TRC105 3 mg/kg Every 2 Weeks | TRC105 10 mg/kg Every 2 Weeks | TRC105 10 mg/kg Weekly | TRC105 15 mg/kg Every 2 Weeks | TRC105 20 mg/kg Every 2 Weeks
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 6 | 4
Participants | 0 | 0 | 0 | 0 | 1 | 0

4. Secondary Outcome: Prostatic-Specific Antigen (PSA) Decline
Description: PSA decline (i.e., PSA greater than 4.0 ng/mL) is defined as two consecutively rising PSA values at a minimum of 1-week intervals (2.0 ng/mL is the minimum starting values for PSA). Normal PSA is 4.0 ng/mL or lower.
Time Frame: 1- week intervals up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | TRC105 1 mg/kg Every 2 Weeks | TRC105 3 mg/kg Every 2 Weeks | TRC105 10 mg/kg Every 2 Weeks | TRC105 10 mg/kg Weekly | TRC105 15 mg/kg Every 2 Weeks | TRC105 20 mg/kg Every 2 Weeks
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 5 | 4
Participants
  PSA Decline >4.0 ng/mL | 0 | 1 | 2 | 2 | 1 | 2
  Normal PSA <4.0 ng/mL | 3 | 2 | 1 | 0 | 4 | 2

5. Secondary Outcome: Clinical Response
Description: Clinical response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response (CR) is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Progressive disease (PD) is at least a 20% decrease in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: 56 days (one cycle = 28 days, restaging post cycle 2)
Measure: Count of Participants; unit: Participants
Arm/Group | TRC105 1 mg/kg Every 2 Weeks | TRC105 3 mg/kg Every 2 Weeks | TRC105 10 mg/kg Every 2 Weeks | TRC105 10 mg/kg Weekly | TRC105 15 mg/kg Every 2 Weeks | TRC105 20 mg/kg Every 2 Weeks
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 6 | 4
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0
  Stable Disease | 3 | 2 | 3 | 2 | 5 | 4
  Progressive Disease | 0 | 1 | 0 | 0 | 0 | 0
  Inevaluable | 0 | 0 | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 43 months, 5 days
Arm/Group | TRC105 1 mg/kg Every 2 Weeks | TRC105 3 mg/kg Every 2 Weeks | TRC105 10 mg/kg Every 2 Weeks | TRC105 10 mg/kg Weekly | TRC105 15 mg/kg Every 2 Weeks | TRC105 20 mg/kg Every 2 Weeks
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/2 | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/3 | 3/3 | 3/3 | 2/2 | 2/6 | 1/4
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 2/2 | 5/6 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRC105 1 mg/kg Every 2 Weeks (N=3) | TRC105 3 mg/kg Every 2 Weeks (N=3) | TRC105 10 mg/kg Every 2 Weeks (N=3) | TRC105 10 mg/kg Weekly (N=2) | TRC105 15 mg/kg Every 2 Weeks (N=6) | TRC105 20 mg/kg Every 2 Weeks (N=4)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0
Infusion related reaction (General disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1 (1) | 1 (1) | 0 | 0 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 (1) | 0 | 0 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 (1) | 0 | 1 (1) | 1 (1) | 1 (1) — Progressive disease
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 2 (2) | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
CPK increased (Investigations) | 0 | 0 | 1 (1) | 0 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Creatinine increased (Investigations) | 0 | 0 | 2 (2) | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 1 (1) | 0 | 0 | 0
Transient ischemic attacks (Nervous system disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1) | 1 (1) | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0
Fever (General disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (2) | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0
Vasovagal reaction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRC105 1 mg/kg Every 2 Weeks (N=3) | TRC105 3 mg/kg Every 2 Weeks (N=3) | TRC105 10 mg/kg Every 2 Weeks (N=3) | TRC105 10 mg/kg Weekly (N=2) | TRC105 15 mg/kg Every 2 Weeks (N=6) | TRC105 20 mg/kg Every 2 Weeks (N=4)
Activated partial thromboplastin time prolonged (Investigations) | 1 (3) | 0 | 1 (1) | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 2 (3) | 2 (2) | 3 (14) | 2 (3) | 2 (5) | 3 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 1 (1) | 1 (1) | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4) | 2 (6) | 0 | 0 | 1 (1)
Chills (General disorders) | 2 (2) | 3 (3) | 1 (2) | 0 | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 0 | 1 (1) | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 | 0 | 0
Creatinine increased (Investigations) | 1 (1) | 0 | 1 (1) | 0 | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 | 1 (1) | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 1 (1) | 0 | 0 | 2 (2)
Edema limbs (General disorders) | 1 (1) | 0 | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (2) | 0 | 1 (1) | 1 (1) | 2 (3)
Fever (General disorders) | 1 (2) | 2 (6) | 3 (13) | 0 | 1 (1) | 2 (4)
Fibrinogen decreased (Investigations) | 1 (2) | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 (1) | 1 (1) | 2 (3) | 0 | 2 (4) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 3 (9) | 1 (1) | 2 (2) | 3 (4) | 3 (4)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 | 0 | 1 (1) | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 (4) | 2 (5) | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 1 (2) | 0 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 | 0 | 0 | 1 (2) | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 | 1 (1) | 0 | 0 | 0
Infusion related reaction (General disorders) | 2 (5) | 1 (1) | 2 (2) | 0 | 0 | 1 (2)
Memory impairment (Nervous system disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 | 0 | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 2 (3) | 2 (5) | 2 (4) | 0 | 0
Pain (General disorders) | 1 (4) | 1 (2) | 2 (2) | 1 (1) | 1 (2) | 2 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 0 | 0 | 0
Renal and urinary disorders - Other, specify (initiating urination) (Renal and urinary disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 (2) | 0 | 1 (1) | 1 (1) | 0 | 0
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 | 1 (1) | 0 | 0 | 0
Weight gain (Investigations) | 1 (1) | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 (2) | 1 (1) | 1 (1) | 0 | 0
Alkaline phosphatase increased (Investigations) | 0 | 1 (2) | 0 | 1 (1) | 1 (1) | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 (1) | 2 (2) | 0 | 0 | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 | 1 (1) | 0 | 0 | 0 | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 0 | 2 (2) | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 1 (2) | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 3 (3) | 1 (1) | 2 (3) | 0 | 0
White blood cell decreased (Investigations) | 0 | 1 (1) | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 (2) | 0 | 0 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 0 | 0 | 0
CPK increased (Investigations) | 0 | 0 | 1 (2) | 0 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 (1) | 0 | 0 | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 (2) | 2 (2) | 4 (7) | 2 (3)
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 (2) | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 0 | 0 | 0
Gastrointestinal disorders - Other, specify (black tarry stools) (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 2 (2) | 0 | 0 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 2 (3) | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1 (1) | 0 | 1 (1) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 2 (2) | 0 | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 2 (3) | 1 (1) | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 1 (2) | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 1 (1) | 0 | 0
Skin and subcutaneous tissue disorders - Other, specify (petechiae) (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Transient ischemic attacks (Nervous system disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Trigeminal nerve disorder (Nervous system disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Weight loss (Investigations) | 0 | 0 | 2 (4) | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (2) | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0
Hot flashes (Vascular disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0
Oral hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1) | 3 (3) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 (1) | 0 | 1 (1)
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 — leg cramping
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 (1) | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 (1)
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1)
Gastrointestinal disorders - Other, specify (gastroenteritis) (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1)
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2012-07-25): https://cdn.clinicaltrials.gov/large-docs/65/NCT01090765/Prot_ICF_000.pdf